CLINICAL TRIAL: NCT06541119
Title: Effect of Selective Strengthening of Peroneus Longus Muscles on Pain Joint Alignment and Foot Function in Hallux Valgus
Brief Title: Effect of Selective Strengthening of Peroneus Longus on Pain , Joint Alignment and Foot Function in Hallux Valgus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Kamel Hassan Alminisi, Senior physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012/005050
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Hallux Valgus
Keywords: Peroneus longus; Hallux valgus angle HVA; Kinovea software; Foot function index; Hallux pain
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sixty mild to moderate Hallux valgus patients will be evaluated for eligibility ; participants will be randomized in 1:1 ratio using computer generated block randomization , followed by concealed allocation by opening quantity numbered sealed envelopes , a card inside will reveal the group assignment as either group A, or group B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective peroneus longus strengthening exercise (Experimental): Group A will receive a weight bearing peroneus longus exercise with conventional physical therapy Programme
  Interventions: Other: Selective Peroneus longus excercise
- Conventional physical therapy programme (Active Comparator): Group B will receive a program consisting of 3 commonly used exercises in Hallux valgus
  Interventions: Other: Conventional physical therapy programme

INTERVENTIONS:
Other: Selective Peroneus longus excercise — Weight bearing peroneus longus exercise
  Other Names: Band heel raises
  Arms: Selective peroneus longus strengthening exercise
Other: Conventional physical therapy programme — * Passive abduction of the Hallux with traction
  * short foot exercise
  * toe spread outs
  Arms: Conventional physical therapy programme

SUMMARY:
Purpose of this study is to measure Change in Hallux valgus angle (HVA )as measured by kinovea software Change in pain as measured by numerical pain rating scale (NPRS) Change in function as measured by Foot function index (FFI )Egyptian version With the peroneus longus strengthening exercise versus the use of conventional physical therapy programme in cases of hallux valgus patients

ELIGIBILITY:
Inclusion Criteria:

* All patients must be diagnosed as having mild to moderate Hallux valgus (with Hallux valgus angle between 15-40 degrees)
* patients aging between 18-60 .
* patients must report pain and limited function .
* patients must report that they are not undergoing physiotherapy , not using orthosis , dynamic splinting exercises for Hallux valgus

Exclusion Criteria:

* Patients diagnosed with systematic diseases such as rheumatoid arthritis .
* Cognitive or mental illness.
* Hallux rigidus or limitus .
* History of surgery to foot of Hallux .
* Previous use of foot orthosis .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Hallux valgus angle HVA | Baseline , 6 weeks (after study completion )
  Hallux valgus angle will be measures musing kinovea software
Level of pain | Baseline , 6 weeks after study completion
  Will be measured using numerical pain rating scale Where 0 represents no pain and 10 represents worst pain imaginable
Foot function | Baseline , 6 weeks after study completion
  Will be measured using Foot Function Index FFI Egyptian version Which is divided into 3 sub categories Pain 0 no pain , 10 worst pain Disability 0 least 10 worst Activity limitation 0 no limitation , 10 worst limitation For the total score, the minimum score is 0% (no pain or difficulty), and maximum score is 100% (worst pain and extreme difficulty requiring assistance).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt